CLINICAL TRIAL: NCT04716179
Title: Prospective Two-arm Study of Fertility in Men With COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Dmitry Enikeev, MD, PhD, Deputy Director for Research, I.M. Sechenov First Moscow State Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: COVID-MFert-20
Record Dates: First submitted 2021-01-17; First posted 2021-01-20 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Covid19; Fertility Issues
MeSH Terms: conditions — COVID-19; Infertility

STUDY DESIGN:
Intervention Model Description: Parallel groups, non-randomized:
  1. - patients with COVID-19;
  2. - healthy participants without COVID-19.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with COVID-19 (Experimental): Patients with confirmed COVID-19 infection
  Interventions: Diagnostic Test: Sperm test; Diagnostic Test: hormone levels (testosterone, FSH, LH, prolactin); Diagnostic Test: SARS-CoV-2 Ig G levels; Other: Testis pathology samples
- Healthy participants (Other): The controlled group with healthy participants without COVID-19 infection.
  Interventions: Diagnostic Test: Sperm test; Diagnostic Test: hormone levels (testosterone, FSH, LH, prolactin); Diagnostic Test: SARS-CoV-2 Ig G levels

INTERVENTIONS:
Diagnostic Test: Sperm test — The semen sample will be collected and analyzed within an hour after collection.
Diagnostic Test: hormone levels (testosterone, FSH, LH, prolactin) — Hormone levels (testosterone, FSH, LH, prolactin) will be assessed on 5-7 days after symptom onset until the end of hospital stay.
Diagnostic Test: SARS-CoV-2 Ig G levels — SARS-CoV-2 Ig G levels will be assessed on 3 months after discharge
Other: Testis pathology samples — Postmortem examination of the testes of patients deceased as a result of COVID-19 infection will be carried out using immunohistochemistry analysis.
  Arms: Patients with COVID-19

SUMMARY:
COVID-19 infection is hypothesized to have a potentially negative effect on male fertility through direct damage to the testes. The current trial is aimed at investigating the effect of SARS-CoV-2 on fertility and determining if viral bodies are capable of directly damaging testicular cells

DETAILED DESCRIPTION:
In late December 2019, the Chinese city of Wuhan witnessed the emergence of a form of pneumonia of unknown etiology. By the middle of January 2020, the disease had managed to spread beyond the country of origin and is now classified by the WHO as the largest pandemic in modern history.

Rapidly spreading and highly contagious, the infection prompted medical professionals all over the world to begin research into the virus with the goal of developing early diagnostic techniques and treatment strategies.

The new pathogen named SARS-Cov-2 belongs to the Coronaviridae family. These viruses cause severe acute respiratory syndrome (SARS-CoV-1, 2002-2003) and Middle East respiratory syndrome (MERS, 2012-2013).

The effects of SARS-CoV-2 on the human body stem from its structure. The spike proteins on the surface of the virus, which are responsible for the name "Coronaviridae," means that it is able to bind to the host receptor protein, angiotensin-converting enzyme 2 (ACE2). This makes cells with high quantities of these receptors on the surface susceptible to the virus.

The genome of SARS-Cov-2 responsible for the COVID-19 pandemic contains both human coronavirus fragments and bat coronavirus fragments (HKU9-1). It is the genetic material of HKU9-1 that makes SARS-CoV-2 unknown to the immune system of the human body.

As of today, three transmission pathways are recognized: close contact, airborne and fomite. Moreover, the virus is known to retain its contagious properties on surfaces for up to 72 hours, and the incubation period ranges between 2 and 14 days. Recent reports indicate that up to 80% of those infected by COVID-19 showed mild or moderate symptoms whereas 20-30% develop severe forms of the disease characterized by shock as well as respiratory and multiple organ failure. According to Chinese and Italian healthcare providers, the mortality rate is between 3.8 and 7.2%.

Zou et al. (2020) reported that non-respiratory symptoms may be explained by the binding of the virus to ACE-2 in other organs. Shen and Wang (2020) proved that ACE-2 is also expressed by testicular cells (namely spermatogonia, Leydig cells and Sertoli cells) which makes them potential targets for the virus. In fact, there are reports of orchitis and epididymitis in patients diagnosed with COVID-19. This means that SARS-CoV-2 may directly damage testicular tissue potentially compromising male fertility.

In a number of studies, PCR did not detect the virus in semen samples obtained during both the acute phase and recovery phase. In another study, postmortem needle and open biopsies of the testicles performed within an hour after death from COVID-19 revealed that testicular tissues were free of SARS-CoV-2 in 10 of 11 cases (91%). At the same time, spermograms in COVID-19 patients showed low ejaculate volume, sperm motility and sperm count. Previously, it was shown that COVID-19 has a severe effect on vasculature and therefore a microthrombi could be a possible contributor to fertility impairment. An assessment of testes with a Doppler enhanced ultrasound was therefore necessary.

Data dedicated to testosterone levels in the blood and inflammatory markers in the semen and testicular tissues is lacking. Available literature indicates changes in the above-mentioned parameters in males with verified COVID-19.

There is ultimately too little information to draw reliable conclusions regarding the effects of the virus on male reproduction. Published reports are limited by small study groups, lack of the control group and absence of follow-up examinations during recovery warranting further research and in-depth exploration of the topic.

ELIGIBILITY:
Inclusion Criteria:

* Clinical or imaging signs of COVID-19 infection
* Nasopharyngeal swab positive for SARS-CoV2 mRNA

Exclusion Criteria:

* Inability to collect semen for analysis
* Congenital anomalies of the testes
* Varicocele
* A history of fertility disorders

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Semen quality analysis - motility | 3 months
  motility of spermatozoa
Semen quantity analysis | 3 months
  count of spermatozoa
Semen quality analysis - shape | 3 months
  shape of spermatozoa

SECONDARY OUTCOMES:
Testosterone | 3 months
  testosteron (ng/dL) level in the blood test
FSH | 3 months
  Follicle-Stimulating Hormone (IU/L) level in the blood test
LH | 3 months
  Luteinizing hormone (IU/L) level in the blood test
Prolactin | 3 months
  prolactin (ng/ml) level in the blood test
Damage of the testes on pathology | 3 months
  Damage of the testes assessment using imminohistochemistry at autopsy specimen

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Enikeev, M.D., Principal Investigator — Sechenov University
Locations (1):
- Sechenov University., Moscow, Russia

IPD SHARING:
Plan to Share IPD: No